CLINICAL TRIAL: NCT02875977
Title: Does a Patient Education Video Augment Pelvic Floor Physical Therapy Compliance?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elizabeth Mueller (Other)
Responsible Party: Sponsor-Investigator, Elizabeth Mueller, MD, Associate Professor, Loyola University
Organization: Loyola University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 208990
Record Dates: First submitted 2016-08-18; First posted 2016-08-23 (Estimated); Results first posted 2018-09-27 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Patient Compliance; Pelvic Floor Disorders
MeSH Terms: conditions — Patient Compliance; Pelvic Floor Disorders

STUDY DESIGN:
Intervention Model Description: Participants are randomized to standard counseling for pelvic floor physical therapy (PFPT) or to an experimental counseling group that comprises both standard counseling and a 4-minute PFPT educational video using a 1:1 allocation
Masking Description: No masking is used in this study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Counseling (Experimental): Patients randomized to this arm receive experimental counseling on the importance of attending PFPT appointments. This includes the standard 2-page educational handout and a 4-minute educational video.
  Interventions: Other: Educational video; Other: Educational handout
- Standard Counseling (Active Comparator): Patients randomized to this arm receive standard counseling on the importance of attending PFPT appointments. This includes the standard 2-page educational handout.
  Interventions: Other: Educational handout

INTERVENTIONS:
Other: Educational video — A 4-minute educational video describing PFPT
  Arms: Experimental Counseling
Other: Educational handout — A 2-page educational handout describing PFPT

SUMMARY:
The investigators intend to measure compliance with attending pelvic floor physical therapy (PFPT) in a Urogynecology population by randomizing patients to either viewing a four minute educational video or reading a handout explaining the therapy.

DETAILED DESCRIPTION:
Patients who have been interviewed, examined, and a plan has been made by the treating physicians in the Female Pelvic Medicine & Reconstructive Surgery practice will be invited to participate at the end of the visit if the patient and physician mutually agree that PFPT is the treatment modality to pursue.

If she agrees to participate, she will be consented and randomized. If she is randomized to standard counseling, she will be given the standard handout to read. If she is randomized to the intervention, she will receive the standard handout and view the 4-minute educational video on an iPad.

At the conclusion of the counseling, patients will be asked if they have any additional questions, and these will be recorded and answered. The patient will also fill out a visual analog scale about how informed she feels regarding PFPT.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have prescribed PFPT by a treating physician in the Female Pelvic Medicine & Reconstructive Surgery practice

Exclusion Criteria:

* Patients ≤ 18 years old

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-08-03 (Actual); Primary Completion 2017-11-15 (Actual); Study Completion 2017-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Brincat, MD, Principal Investigator — Loyola University; Elizabeth Mueller, MD, Study Director — Loyola University
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data with other researchers

REFERENCES:
- [Background] Dumoulin C, Alewijnse D, Bo K, Hagen S, Stark D, Van Kampen M, Herbert J, Hay-Smith J, Frawley H, McClurg D, Dean S. Pelvic-Floor-Muscle Training Adherence: Tools, Measurements and Strategies-2011 ICS State-of-the-Science Seminar Research Paper II of IV. Neurourol Urodyn. 2015 Sep;34(7):615-21. doi: 10.1002/nau.22794. Epub 2015 May 21. PMID 25998493
- [Background] Fitzgerald MP, Anderson RU, Potts J, Payne CK, Peters KM, Clemens JQ, Kotarinos R, Fraser L, Cosby A, Fortman C, Neville C, Badillo S, Odabachian L, Sanfield A, O'Dougherty B, Halle-Podell R, Cen L, Chuai S, Landis JR, Mickelberg K, Barrell T, Kusek JW, Nyberg LM; Urological Pelvic Pain Collaborative Research Network. Randomized multicenter feasibility trial of myofascial physical therapy for the treatment of urological chronic pelvic pain syndromes. J Urol. 2013 Jan;189(1 Suppl):S75-85. doi: 10.1016/j.juro.2012.11.018. PMID 23234638
- [Background] Alewijnse D, Mesters I, Metsemakers J, Adriaans J, van den Borne B. Predictors of intention to adhere to physiotherapy among women with urinary incontinence. Health Educ Res. 2001 Apr;16(2):173-86. doi: 10.1093/her/16.2.173. PMID 11345660
- [Background] Tibaek S, Dehlendorff C. Do women with pelvic floor dysfunction referred by gynaecologists and urologists at hospitals complete a pelvic floor muscle training programme? A retrospective study, 1992-2008. Int Urogynecol J. 2013 Aug;24(8):1361-9. doi: 10.1007/s00192-012-2018-2. Epub 2013 Jan 5. PMID 23291858
- [Derived] Shannon MB, Adams W, Fitzgerald CM, Mueller ER, Brubaker L, Brincat C. Does Patient Education Augment Pelvic Floor Physical Therapy Preparedness and Attendance? A Randomized Controlled Trial. Female Pelvic Med Reconstr Surg. 2018 Mar/Apr;24(2):155-160. doi: 10.1097/SPV.0000000000000516. PMID 29474290

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from August 2016 through March 2017 (7 months) from a tertiary care female pelvic medicine and reconstructive surgery practice.
Groups:
- Experimental Counseling: Patients randomized to this arm receive experimental counseling on the importance of attending pelvic floor physical therapy (PFPT) appointments. This includes the standard 2-page educational handout and a 4-minute educational video.
Period: Overall Study
Arm/Group | Experimental Counseling | Standard Counseling
Started | 100 | 100
Completed | 58 | 71
Not Completed | 42 | 29
Not completed — Lost to Follow-up | 42 | 29

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Counseling | Standard Counseling | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.32 (16.12) | 56.77 (17.00) | 57.05 (16.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 100 | 200
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 24 | 48
  Not Hispanic or Latino | 76 | 75 | 151
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 13 | 28
  White | 81 | 78 | 159
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 2 | 6 | 8
Region of Enrollment [Number; unit: participants]
  United States | 100 | 100 | 200
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 32.48 (8.24) | 29.94 (6.74) | 31.21 (7.62)
Primary Language [Count of Participants; unit: Participants]
  English | 95 | 94 | 189
  Spanish | 5 | 6 | 11
Vaginal Parity [Median (Inter-Quartile Range); unit: Pregnancies to a viable gestational age] | 2 [1 to 3] | 2 [1 to 3] | 2 [1 to 3]
Urogynecologic diagnosis [Count of Participants; unit: Participants]
  Stress Urinary Incontinence (SUI) | 9 | 25 | 34
  Urgency Urinary Incontinence (UUI) | 25 | 24 | 49
  Mixed Urinary Incontinence (MUI) | 34 | 21 | 55
  Urgency-frequency syndrome | 27 | 20 | 47
  Weak Pelvic Floor | 8 | 14 | 22
  Defecatory dysfunction | 6 | 6 | 12
  Pelvic Organ Prolapse (POP) | 10 | 12 | 22
  Myofascial Pain | 40 | 36 | 76
  Other Urogynecologic Diagnosis | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Completed PT Visits
Description: The number of patients who completed at least half of their recommended PFPT visits is compared between those assigned to enhanced counseling versus standard counseling
Time Frame: 3 months
Population: This analysis comprises only the participants who were randomized and had follow-up PFPT completion information available
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Counseling | Standard Counseling
Number analyzed (Participants) | 58 | 71
Participants
  Completed half of the recommended visits | 47 | 50
  Did not complete half of the recommended visits | 11 | 21
Statistical Analysis 1: Comparison: Experimental Counseling vs Standard Counseling; The null hypothesis is that there is no difference in the odds of completing half of the recommended PFPT visits between those assigned to standard versus experimental counseling; Test type: Superiority; p = 0.17, Regression, Logistic; Odds Ratio (OR) = 1.794, 95% CI 2-sided [0.782 to 4.119]

2. Secondary Outcome: Initiation of PFPT
Description: The number of patients who initiated PFPT is compared between those assigned to enhanced counseling versus standard counseling
Time Frame: 3 months
Population: This analysis comprises all participants who were randomized
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Counseling | Standard Counseling
Number analyzed (Participants) | 100 | 100
Participants
  Initiated PFPT | 58 | 71
  Did not initiate PFPT | 42 | 29
Statistical Analysis 1: Comparison: Experimental Counseling vs Standard Counseling; The null hypothesis is that there is no difference in the odds of initiating PFPT between those assigned to standard versus experimental counseling; Test type: Superiority; p = 0.056, Regression, Logistic; Odds Ratio (OR) = 0.564, 95% CI 2-sided [0.314 to 1.014]

3. Secondary Outcome: PFPT Discharge
Description: The number of patients who discharged from PFPT is compared between those assigned to enhanced counseling versus standard counseling
Time Frame: 3 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Counseling | Standard Counseling
Number analyzed (Participants) | 58 | 71
Participants
  Discharged from PFPT | 27 | 33
  Not discharged from PFPT | 29 | 37
  PFPT discharge status unknown | 2 | 1
Statistical Analysis 1: Comparison: Experimental Counseling vs Standard Counseling; The null hypothesis is that there is no difference in the odds of discharge from PFPT between those assigned to standard versus experimental counseling; Test type: Superiority; p = 0.90, Regression, Logistic; The statistical test of the hypothesis excludes the three individuals with unknown PFPT discharge status; Odds Ratio (OR) = 1.044, 95% CI 2-sided [0.517 to 2.110]

4. Secondary Outcome: Days to Initiation of PFPT
Description: The number of days from referral to PFPT to the first PFPT visit is compared between those assigned to enhanced counseling versus standard counseling
Time Frame: 3 months
Population: This analysis comprises only the participants who were randomized and initiated PFPT
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Experimental Counseling | Standard Counseling
Number analyzed (Participants) | 58 | 71
Days | 15 [7 to 23] | 19 [11 to 31]
Statistical Analysis 1: Comparison: Experimental Counseling vs Standard Counseling; Among those who initiated PFPT therapy, the null hypothesis is that there is no difference in the number of days to initiating PFPT therapy between those assigned to standard versus experimental counseling; Test type: Superiority; p = 0.16, Wilcoxon (Mann-Whitney); Z-Score = -1.4262

5. Secondary Outcome: Change in Urogenital Distress From Baseline to 3 Months
Description: Patients complete the Urinary Distress Inventory 6 (UDI-6) prior to beginning PFPT therapy and following PFPT therapy. The change in UDI-6 from baseline to 3 months following therapy is compared between those assigned to enhanced counseling versus standard counseling. The UDI-6 is an assessment of urogenital distress with a score range from 0 to 100, where higher scores indicate greater disability.
Time Frame: 3 months
Population: This analysis comprises only the participants who were randomized and had pre-PFPT and post-PFPT UDI-6 scores available
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental Counseling | Standard Counseling
Number analyzed (Participants) | 27 | 24
units on a scale | -12.04 (21.29) | -16.49 (25.46)
Statistical Analysis 1: Comparison: Experimental Counseling vs Standard Counseling; The null hypothesis is that there is no difference in the change from pre-PFPT to post-PFPT UDI-6 scores between those assigned to standard versus experimental counseling; Test type: Superiority; p = 0.50, t-test, 2 sided; Mean Difference (Final Values) = -4.456, 95% CI 2-sided [-17.6149 to 8.7028], Standard Error of Mean 6.5481

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 11 months
Arm/Group | Experimental Counseling | Standard Counseling
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 0/100 | 0/100

LIMITATIONS AND CAVEATS:
There are no limitations or caveats to report

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-01): https://cdn.clinicaltrials.gov/large-docs/77/NCT02875977/Prot_SAP_000.pdf